CLINICAL TRIAL: NCT04411485
Title: Evaluation of Sexual Satisfaction and Sexual Dysfunction in Partner of Patients With Ankylosing Spondylitis
Brief Title: Sexual Dysfunction in Partner of Patients With Ankylosing Spondylitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Ayan, Principal Investigator, Antalya Training and Research Hospital
Other Study IDs: 2016-098
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Ankylosing Spondylitis; Sexual Dysfunction
Keywords: Ankylosing spondylitis; sexual dysfunction
MeSH Terms: conditions — Spondylitis, Ankylosing; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of Ankylosing Spondylitis: Patient with ankylosing spondylitis diagnosed by a rheumatologist
  Interventions: Other: Sexual dysfunction
- Group of control: Healthy volunteers of the same age and gender as patients
  Interventions: Other: Sexual dysfunction

INTERVENTIONS:
Other: Sexual dysfunction — Sexual dysfunction will be determined with separate scales for women and men

SUMMARY:
The adverse effects of rheumatologic diseases, especially Ankylosing Spondylitis (AS), on sexual functions are known. The causes of sexual dysfunction in rheumatologic diseases are due to factors such as pain, weakness, fatigue, stiffness, functional disability, anxiety, depression, hormonal deficiency, drug use, decreased libido and poor body image. Depending on these factors, sexual intercourse and frequency of sexual intercourse may decrease. Sexual dysfunction may be seen in AS due to physical and emotional problems caused by the disease.

DETAILED DESCRIPTION:
There are many studies in the literature that determine sexual satisfaction and sexual dysfunction in individuals with AS and compare individuals with AS to healthy individuals . In the light of these studies, the investigators thought that the sexual function of partner of individuals with AS may also be affected negatively. In the literature, no previous study examines the sexual function of partner of individuals with AS. Therefore, the aim was to determine the sexual function of partner of individuals with AS and to compare with healthly adults of the same sex.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with AS for individuals with AS,
* No additional disease (comorbid and psychiatric disease, hypothyroidism, hypopituitarism, hypogonadism or hyperprolactinemia)
* Having a partner (relationship status in a monogamous sexual relationship),
* Not smoking and drinking,
* Non-AS partner have not been diagnosed with AS and their partner is AS.

Exclusion Criteria:

* Overweight or obesity (BMI <28 kg / m2)
* Having had a pelvic injury, urological or gynecological operation in the last 3 months
* Hypogonadism; penile abnormalities such as hypospadias, congenital curvature or Peyronie's disease with preserved penis stiffness
* Prostatic disorder
* Use of drugs that may affect erectile function (steroids, antihistamines, ß-blockers or SSRIs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ankylosing spondylitis diagnosed by the rheumatologist
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Scale | 1 week
  It is a Likert-type scale that evaluates sexual dysfunction in women consisting of 19 items. The validity and reliability study of FSFI was performed by Rosen et al. (8). The scale consists of six items: desire, arousal, lubrication, orgasm, sexual satisfaction and pain. Each title is scored between 0 or 1 to 6. The lowest score is two (2) and the highest score is thirty-six (36). A higher score means better function. Rosen et al. (2000) in their study of functional status; The FSFI score was classified as good if> 30, moderate between 23-29, and poor if <23 .
International Erectile Function Form | 1 week
  The questionnaire, which consists of 15 questions in total, determines the participants' erectile function, orgasmic function, sexual desire, sexual satisfaction and overall satisfaction and these 5 different sexual function areas are scored according to the answers received. It is a Likert type scale. As the score increases, it means that each area is good.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Tarining and Research Hospital Ethics Commitee, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is a data to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Liu YF, Dong H, Chen Z, Wang YU, Tu SH. Impact of ankylosing spondylitis on sexual function: A systematic review and meta-analysis. Exp Ther Med. 2015 Apr;9(4):1501-1507. doi: 10.3892/etm.2015.2239. Epub 2015 Jan 29. PMID 25780459